CLINICAL TRIAL: NCT01155765
Title: Prasugrel in Comparison to High Clopidogrel Dose for Inhibition of Platelet Reactivity as Assessed With a Point-of-Care Platelet Function Assay in Patients Undergoing Chronic Hemodialysis Presenting Resistance to the Usual Clopidogrel Dose
Brief Title: Prasugrel Versus High Dose Clopidogrel in Clopidogrel Resistant Patients Undergoing Chronic Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Dimitrios Alexopoulos, Patras University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PATRASCARDIOLOGY-2
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-04

CONDITIONS: Hemodialysis; Chronic Renal Failure
Keywords: Clopidogrel Resistance; prasugrel; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prasugrel (Experimental): Prasugrel per os 10 mg/day
  Interventions: Drug: Prasugrel
- Clopidogrel (Active Comparator): Clopidogrel per os 150 mg/day
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Prasugrel — Prasugrel 10 mg/day for 15 days
  Arms: Prasugrel
Drug: Clopidogrel — Clopidogrel 150 mg/day for 15 days
  Arms: Clopidogrel

SUMMARY:
Clopidogrel administration is essential in patients undergoing percutaneous coronary intervention, in patients with previous stroke, in patients under chronic hemodialysis via fistulae and in patients with chronic atrial fibrillation if coumarin administration is not a viable option. Patients with chronic renal failure present lower clopidogrel response compared to those with normal renal function. Additionally, hemodialysis via the dialysis filter causes a decrease in glycoprotein platelet receptors, potentially associated with thienopyridine hyporesponsiveness. Clopidogrel resistant patients as assessed by VerifyNow P2Y12(Accumetrics)will be randomized in 1:1 fashion to prasugrel 10mg/day or clopidogrel 150mg/day. On day 15±2 days a crossover directly to the alternate treatment group will be carried out, without an interventing washout period. All patients will undergo platelet reactivity assessment, documentation of major adverse cardiac events and documentation of any serious adverse events(stroke, bleeding)at day 15 and day 30.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. History of chronic renal failure under hemodialysis for at least 6 months
3. Under clopidogrel 75mg/day treatment for at least 7 days before randomization
4. Informed consent obtained in writing

Exclusion Criteria:

1. Treatment with other investigational agents (including placebo) or devices within 30 days prior to randomization or planned use of investigational agents or devices prior to the Day 30 visit.
2. Pregnancy
3. Breastfeeding
4. Inability to give informed consent or high likelihood of being unavailable for the Day 30 follow up.
5. Malignancy
6. Acute coronary syndrome or hemodynamic instability within 30 days prior to randomization
7. Requirement for oral anticoagulant prior to the Day 30 visit
8. Requirement for discontinuation of thienopyridine treatment prior to the Day 30 visit
9. Treatment with IIb/IIIa inhibitors within 30 days prior to randomization or planned administration prior to the Day 30 visit
10. Known hypersensitivity to prasugrel or clopidogrel.
11. History of gastrointestinal bleeding, genitourinary bleeding or other site abnormal bleeding within the previous 6 months.
12. Other bleeding diathesis, or considered by investigator to be at high risk for bleeding on thienopyridine therapy.
13. Any previous history of ischemic stroke, intracranial hemorrhage or disease (neoplasm, arteriovenous malformation, aneurysm).
14. Thrombocytopenia (<100.000 / μL) at randomization
15. Known liver failure (bilirubin > 2mg/dl)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Platelet Reactivity Units (PRU)assessed by VerifyNow P2Y12(Accumetrics) | Day 30

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (death, myocardial infarction, revascularization) | Day 30
Hemorrhage | Day 30
Stroke | Day 30

CONTACTS AND LOCATIONS:
Locations (1):
- Patras University Hospital, Pátrai, Achaia, Greece

REFERENCES:
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730